CLINICAL TRIAL: NCT07035366
Title: Two Procedures for Uniportal Video Assisted Thoracoscopic Surgery to Treat Severe Cases of Diaphragmatic Eventration in Adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Dina Mohamed Osman, assisstant professor, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZU-IRB # 738/15-oct-2024
Record Dates: First submitted 2025-06-12; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Diaphragmatic Eventration
Keywords: stabled resection; running sutures; diaphragmatic eventration
MeSH Terms: conditions — Diaphragmatic Eventration

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- running sutures (Experimental): diaphragmatic plication by running sutures
  Interventions: Procedure: running sutures
- stabled resection (Experimental): diaphragmatic plication by stabled resection
  Interventions: Procedure: stabled resection

INTERVENTIONS:
Procedure: stabled resection — diaphragmatic plication of sever eventration by stabled resection
  Arms: stabled resection
Procedure: running sutures — plication of diaphragmatic eventration by running sutures
  Arms: running sutures

SUMMARY:
highly elevated abnormal diaphragm is lowered to normal position by runuing suture accordion shaped or cut part of diphragm by stabler

DETAILED DESCRIPTION:
high degree of eventration is corrected either stabled resection or running sutures

ELIGIBILITY:
Inclusion Criteria:

* patients who presented with dyspnea or orthopnea with sever eventration

Exclusion Criteria:

* other causes of dyspnea or elevated hemidiaphragm

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2024-12-10 (Actual); Study Completion 2025-03-15 (Actual)

PRIMARY OUTCOMES:
Cosmetic & Recovery Time (days) | 1 week after surgery
operative time (min) | from the start of skin incision till the extubation of the patient
postoperative pain(pain score) | postoperative pain recieved by operated patient
lung function recovery (lung function test) | lung function test done one and three months postoperative
  forced expiratory volume in 1st second,

CONTACTS AND LOCATIONS:
Locations (3):
- Egypt (3):
  - cardiothoracic surgery department-faculty of medecine-Zagazig univeristy-Egypt, Zagazig, Sharqia Province
  - cardiothorathic surgery department -faculty of medecine-zagazig univeristy-Egypt, Zagazig, Sharqia Province
  - Cardiothoracic Surgery Department-Faculty of Mdecine-Zagazig Univeristy, Zagazig, Sharqia Province

IPD SHARING:
Plan to Share IPD: No